CLINICAL TRIAL: NCT04181177
Title: Randomized, Comparative Study to Evaluate the Effects of Cosmetic Balm on Xerosis and Associated Signs and Symptoms, Induced by Systemic Anticancer Treatments in Subjects Receiving Targeted Educational Action Compared to a Control Group
Brief Title: Efficacy Study of Cosmetic Product on Xerosis Induced by Systemic Anticancer Treatments
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV4429A2018386
Record Dates: First submitted 2019-11-20; First posted 2019-11-29 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Xerosis
Keywords: anticancer treatment; targeted educational action; pruritus; quality of life; NCI CTCAE; Patient Global Assessment; Investigator Global Assessment; Dermatology Life Quality Index (DLQI); Hydration Index (HI); Numeric Scale (NS)
MeSH Terms: conditions — Pruritus | interventions — Cosmetics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Informed group: This group will receive the Cosmetic product RV4429A balm and targeted educational action between V1 and V2 or between V2 and V3 according to the randomization
  Interventions: Other: Cosmetic product
- Control group: The control group, in the first period between V1 and V2, is a group not informed about his skin condition, not receiving any emollient product and not receiving targeted educational action. It's representative of the real life called "best supportive care/Supportive care": the doctor prescribes what it seems to be the best for his patient according to his opinion in view of his condition, at a given moment.
  A high variability exists within this group. In order to answer the investigator's hypothesis and demonstrate the effectiveness of the RV4429A balm, the parallel group design is chosen for the first follow-up period and then a second follow-up period is chosen for the initial control group to replace the inter-individual variability by intra-individual variability.

INTERVENTIONS:
Other: Cosmetic product — Cosmetic balm: application twice daily on the whole body in sufficient quantity to cover all the xerosis areas. It contains an I-modulia(r) complex which decreases the sensation of itching, CER-OMEGA which are lipids similar to those of the skin, help repair and nourish the skin, finally Avène Thermal Spring Water which have soothing and softening properties.
  Targeted education action consist in advices and preventive measures (including hygiene) regarding xerosis and associated dermatological signs / symptoms. Emollient and application tips and other supportive care tips will be provided. The targeted educational action will be monitored by the medical and paramedical teams (specialized nurses).
  Groups: Informed group

SUMMARY:
Xerosis is one of the most common adverse events in patients treated with new cancer therapies and chemotherapies, such as multi-kinase inhibitors and more specifically, immunological checkpoint inhibitors used in the treatment of several cancers.

Xerosis appears as a result of a deterioration of the stratum corneum which results in a reduction of the hydric power of the skin. It reaches the trunk and limbs, with an incidence of 4-35%, and gradually disappears after the end of treatment.

Preventive targeted educational action is essential before initiation of cancer treatment. Once the xerosis is installed, the management is based on the use of emollients to contribute to the hydric correction of the skin. In the case of inflammation or associated infection, the administration of topical corticosteroids and / or local or oral antibiotic therapy is prescribed.

The aim of this study is to evaluate the efficacy of the cosmetic product (balm) on the improvement of xerosis induced by systemic anticancer treatments, in participants receiving targeted educational action compared to a control group.

Clinical, biological and biometrological assessments will be performed to characterized the effects in both induced xerosis and associated signs and symptoms.

Each group will include 40 participants.

DETAILED DESCRIPTION:
Systemic anticancer treatments, whether they are conventional molecules or more current molecules such as targeted therapies, are responsible for numerous dermatological adverse effects, notably xerosis, the repercussions of which may lead to a decrease in compliance, dose reductions or even a complete cessation of cancer treatment.

To date, the management of these adverse effects is not performed routinely and published efficacy data on secondary side effects are missing.

The purpose of this comparative study is to evaluate the clinical efficacy of the RV4429A balm combined with a targeted educational action, on the improvement of induced xerosis on the one hand and on the improvement of the signs and symptoms associated with this induced xerosis. on the other hand ; based on clinical, biometrological and biological criteria. The objective is to provide data on this product in this symptomatology.

Xerosis and the associated dermatological signs / symptoms will be assessed individually as well as through overall scores, as measured by both the investigator and the patient as clinical expression is often poorly correlated with psychic and functional impact. Quality of life, cosmetic acceptability and targeted educational action and tolerance will also be assessed.

The improvement of the quality of life of the patients, the reduction of the undesirable effects induced could thus guarantee the observance of the patients vis-à-vis the anticancer treatments.

The study area is the whole body. A target area will be chosen and will be located on one of the upper limbs (outside the hands) or on the trunk (outside a hairy area). The target area is defined as the xerosis area representative of the the most severe xerotic state, according to the investigator's opinion.

The dermatologist who will evaluate the participant should be, as far as possible, the same throughout the study.

A second period will be carried out by the participants of the control group who will enter in the targeted educational action phase of in their turn.

The study includes 2 visits for the informed group and 3 visits for the control group:

* V1 (J1) - Inclusion (common to both groups)
* V2 (J21 ± 2J or J28 ± 2J) - End of study (informed group) - Intermediate (control group)
* V3 (J42 ± 2J or J56 ± 2J) - End of study (control group) The dates of the visits 2 and 3 will be adapted to the frequency of the visits of administration of the anticancer treatment.

The maximum duration of participation for a participant may be 23 days or 44 days or it may be 30 days or 58 days from the inclusion visit to the end-of-study visit, depending on the group and depending the timeframe between cancer treatment visits.

All subjects in the control group will enter onto the informed group after three weeks or one month (depending on the timeframe between cancer treatment visits), regardless of their condition (presence or absence of on-going xerosis).

ELIGIBILITY:
Inclusion Criteria:

1. Criteria related to the population:

   * Subject having signed his/her written informed consent for his/her participation in the study
   * Subject affiliated to a social security system or health insurance, or is a beneficiary
   * Subject with phototype I, II, III, IV according to the Fitzpatrick scale
   * For woman of childbearing potential: use of an effective method of contraception, as assessed by the investigator for at least 4 weeks before inclusion in the study and using it during the whole duration of the study
2. Criteria related to diseases and general health:

   * Subject having a grade ≥ 2 of dry skin on NCI-CTCAE scale in 3 grades, assessed on the entire body
   * Subject having an intensity of dry skin ≥ 3, according a 5-points scale, on the target area
   * Subject having a general state of clinical and/or physical health adequate(s) to carry out the study according to the investigator's opinion, and presenting a total score ≤ 1 according to the "performance status" scale of WHO (World Health Organization) in 5-points
3. Criteria related to treatments:

   * On-going systemic anticancer treatment, whatever the dosage and whatever the duration of treatment

Exclusion Criteria:

1. Criteria related to the population:

   * For woman of childbearing potential: pregnant or breastfeeding or planning to be pregnant during the study
   * Subject unable to understand the information given including study procedures (for linguistic or psychiatric reasons) and to give his/her consent in writing
   * Subject who, in the judgement of the investigator, is not likely to be compliant during the study
   * Subject who has forfeited his/her freedom by administrative or legal award or is under guardianship
   * Subject is in a position likely to represent a conflict of interest and/or is a family member of any people involved in the conduct of the study (secretary, nurse, technician,…), of the investigational site
   * Subject who is currently participating, who plans to participate or who has participated within the previous weeks in another clinical study liable to interfere with the study assessments according to the investigator's assessment
   * Subject unable to write required information in a subject diary
2. Criteria related to diseases and general health

   * Subject having a grade= 3 of pruritus on NCI-CTCAE scale in 3 grades, assessed on the entire body
   * Subject presenting infectious (viral, bacterial, fungal) or inflammatory complications, on the entire body
   * Subject with a history of atopic or contact dermatitis
   * Subject presenting any other dermatological condition the day of the visit (atopic or contact dermatitis, chronic xerosis, ..), liable to interfere with the study assessments, according to the investigator's opinion
   * Subject with history of allergy or intolerance to any of the study products ingredients
3. Criteria related to treatments and cosmetic products

   * Radiotherapy in progress or planned during the study
   * Application of dermocorticoïdes during 5 consecutive days within the 10 days previous the visit
   * Any other topical or systemic treatment previously used or on-going (other than systemic anticancer treatment and antihistaminic) liable to interfere with the study assessments or incompatible with the study procedures, according to the investigator's opinion
   * Application of any other topical treatment or topical cosmetic product (except hygiene product), liable to interfere with the study assessments, according to the investigator's opinion, on the entire body, the day of the visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are selected during their usual medical care with their oncologist in the investigational site.
  Subjects The subjects corresponding to eligibility criteria may receive a phone call, a letter or an e-mail proposing to participate to the study.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
dry skin on scale NCI CTCAE 5.0 | Change from baseline to 3 weeks or 4 weeks later according to the frequency of participant's oncologic received treatment, for each group, on the entire body
  * Grade1: Covering <10% BSA* and no associated erythema or pruritus
  * Grade2: Covering 10 - 30% BSA* and associated with erythema or pruritus; limiting instrumental ADL*
  * Grade3: Covering >30% BSA* and associated with pruritus; limiting self care ADL* * BSA : Body Surface Area, ADL : Activities of Daily Living

SECONDARY OUTCOMES:
dry skin on scale NCI CTCAE 5.0 | Day 21 or Day 28 (according to the frequency of participant's oncologic received treatment) and Day 42 or Day 56 (according to the frequency of participant's oncologic received treatment), for group control, on the entire body
  * Grade1: Covering <10% BSA* and no associated erythema or pruritus
  * Grade2: Covering 10 - 30% BSA* and associated with erythema or pruritus; limiting instrumental ADL*
  * Grade3: Covering >30% BSA* and associated with pruritus; limiting self care ADL* * BSA : Body Surface Area, ADL : Activities of Daily Living
pruritus on scale NCI CTCAE 5.0 | Change from baseline to 3 weeks or 4 weeks later according to the frequency of participant's oncologic received treatment, for each group, on the entire body
  * Grade1: Mild or localized; topical intervention indicated
  * Grade2: Widespread and intermittent; skin changes from scratching (e.g., edema, papulation, excoriations, lichenification, oozing/crusts); oral intervention indicated; limiting instrumental ADL
  * Grade3: Widespread and constant; limiting self care ADL or sleep; systemic corticosteroid or immunosuppressive therapy indicated
pruritus on scale NCI CTCAE 5.0 | Day 21 or Day 28 (according to the frequency of participant's oncologic received treatment) and Day 42 or Day 56 (according to the frequency of participant's oncologic received treatment), for each group, on the entire body
  * Grade1: Mild or localized; topical intervention indicated
  * Grade2: Widespread and intermittent; skin changes from scratching (e.g., edema, papulation, excoriations, lichenification, oozing/crusts); oral intervention indicated; limiting instrumental ADL
  * Grade3: Widespread and constant; limiting self care ADL or sleep; systemic corticosteroid or immunosuppressive therapy indicated
dry skin on 5-points scale | Change from baseline to 3 weeks or 4 weeks later according to the frequency of participant's oncologic received treatment, for each group, on the target area
  0: absent; 1: very mild; 2: mild; 3: moderate; 4: severe
dry skin on 5-points scale | Day 21 or Day 28 (according to the frequency of participant's oncologic received treatment) and Day 42 or Day 56 (according to the frequency of participant's oncologic received treatment), for each group, on the target area
  0: absent; 1: very mild; 2: mild; 3: moderate; 4: severe
Investigator Global Assessment (IGA) on 5-points scale | Day 21 or Day 28 (according to the frequency of participant's oncologic received treatment) and Day 42 or Day 56 (according to the frequency of participant's oncologic received treatment), for each group, on the target area
  0: aggravation; 1: no change; 2: slight improvement; 3: clear improvement; 4: total improvement
Patient Global Assessment (PGA) on 5-points scale | once a week at home (before application if any), during 3 weeks or 4 weeks according to the frequency of participant's oncologic received treatment, for informed group, on the target area
  0: aggravation; 1: no change; 2: slight improvement; 3: clear improvement; 4: total improvement
Patient Global Assessment (PGA) on 5-points scale | once a week at home (before application if any), during 6 weeks or 8 weeks according to the frequency of participant's oncologic received treatment, for control group, on the target area
  0: aggravation; 1: no change; 2: slight improvement; 3: clear improvement; 4: total improvement
dryness/tightness; tingling; warming/burning; pruritus/itching; discomfort | once a week at home (before application if any), during 3 weeks or 4 weeks according to the frequency of participant's oncologic received treatment, for informed group, on the target area
  Numeric Scale 0-10
dryness/tightness; tingling; warming/burning; pruritus/itching; discomfort | once a week at home (before application if any), during 6 weeks or 8 weeks according to the frequency of participant's oncologic received treatment, for control group, on the target area
  Numeric Scale 0-10
Dermatology Life Quality Index questionnaire (DLQI) | Change from baseline to 3 weeks or 4 weeks later according to the frequency of participant's oncologic received treatment, for each group
  Questionnaire Score 0-30
Dermatology Life Quality Index questionnaire (DLQI) | Day 21 or Day 28 (according to the frequency of participant's oncologic received treatment) and Day 42 or Day 56 (according to the frequency of participant's oncologic received treatment), for each group
  Questionnaire Score 0-30
Cosmetic acceptability questionnaire | 3 weeks or 4 weeks according to the frequency of participant's oncologic received treatment, for informed group
  Questionnaire ad-hoc
Cosmetic acceptability questionnaire | 6 weeks or 8 weeks according to the frequency of participant's oncologic received treatment, for control group
  Questionnaire ad-hoc
Targeted educational action questionnaire | 3 weeks or 4 weeks according to the frequency of participant's oncologic received treatment, for informed group
  Questionnaire ad-hoc
Targeted educational action questionnaire | 6 weeks or 8 weeks according to the frequency of participant's oncologic received treatment, for control group
  Questionnaire ad-hoc
Hydration Index (IH) | Change from baseline to 3 weeks or 4 weeks later according to the frequency of participant's oncologic received treatment, for each group, on target area
  Measure by corneometer
Hydration Index (IH) | Day 21 or Day 28 (according to the frequency of participant's oncologic received treatment) and Day 42 or Day 56 (according to the frequency of participant's oncologic received treatment), for each group, on target area
  Measure by corneometer
Corneocytes quantification | Change from baseline to 3 weeks or 4 weeks later according to the frequency of participant's oncologic received treatment, for each group, on target area
  Sampling performed with DSquame disc and image taking with C-Cube probe.
Corneocytes quantification | Day 21 or Day 28 (according to the frequency of participant's oncologic received treatment) and Day 42 or Day 56 (according to the frequency of participant's oncologic received treatment), for each group, on target area
  Sampling performed with DSquame disc and image taking with C-Cube probe.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent SIBAUD, Dr, Principal Investigator — Institut Universitaire du Cancer Toulouse- Oncopole
Locations (4):
- France (4):
  - Centre Hospitalier de Cahors, Cahors
  - Centre Hospitalier de Carcassonne, Carcassonne
  - Centre Hospitalier de Tarbes, Tarbes
  - Institut Universitaire du Cancer Toulouse- Oncopole, Toulouse

IPD SHARING:
Plan to Share IPD: No